CLINICAL TRIAL: NCT05040867
Title: Effects of Physical Exercise, and Its Prescription Guided by Heart Rate Variability, on the Cardiotoxicity, Physical and Psychological Health of Breast Cancer Patients
Brief Title: Exercise Prescription Guided by Heart Rate Variability in Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GO fit Lab- Ingesport (Network)
Collaborators: Marqués de Valdecilla University Hospital (Unknown); Center for Sport Studies, Rey Juan Carlos University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CARDIEJERCAN
Record Dates: First submitted 2021-08-24; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer; Cardiotoxicity; Autonomic Imbalance
Keywords: Physical exercise; Heart rate variability; Strength training; Cardiovascular training; Cardiotoxicity changes; Cancer patients; Cancer-related side effects; High-intensity training
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (CG) (No Intervention): Participants will continue with their daily life and usual care.
- Traditional periodization exercise group (TEG) (Experimental): Participants will participate in a physical exercise program with a preplanned intensity progression.
  Interventions: Other: Physical exercise program
- Heart Rate Variability exercise group (HRVG) (Experimental): Participants will participate in a physical exercise program guide by participants' daily heart rate variability to plan the intensity progression.
  Interventions: Other: Physical exercise program

INTERVENTIONS:
Other: Physical exercise program — The physical exercise programme will last 16 weeks where participants will do three weekly sessions of 60 minutes, approximately. In these training sessions, cardiovascular and strength components will be worked out, planned from moderate to high intensity in the TEG and unique high intensity in the HRVG. The training programme will be divided into three mesocycles from neuromuscular adaptation to reach, in last period, the highest loads and cardiovascular levels. Each session will include a warm-up, a main part and a cool-down with stretching and mobility exercises.
  The difference between the interventions of the HRVG and TEG will be in the planning of the intensity of the cardiovascular exercises and the weight to be lifted in the strength exercises. The first session of both programmes will have the same intensity but depending on how the heart rate variability of the HRVG patients reacts to, the weight and the intensity will be individualised each day.
  Arms: Heart Rate Variability exercise group (HRVG); Traditional periodization exercise group (TEG)

SUMMARY:
Breast cancer is a chronic disease that has seen a boom in research into its treatments, improvements and effects in recent decades. These advances have also highlighted the need to use physical exercise as a countermeasure to reduce the cardiotoxicity of pharmacological treatments. Patients need a correct daily individualisation of the exercise dose necessary to produce the physiological, physical and psychological benefits. To this end, the present study will use, in a novel way in this population, heart rate variability (HRV) as a measure of training prescription. The primary objective of this randomised clinical trial is to analyse the effects of a physical exercise programme planned according to daily HRV in breast cancer patients after chemotherapy treatment. For this purpose, a 16-week intervention will be carried out with 90 breast cancer patients distributed in 3 groups (control group, conventional preprogrammed physical exercise training group and physical exercise group with HRV daily programming). Cardiorespiratory capacity, strength, flexibility, agility, balance, body composition, quality of life, fatigue, functionality, self-esteem, anxiety and depression of patients before and after the intervention will be evaluated in order to compare the effects of exercise and its programming.

DETAILED DESCRIPTION:
The intervention of 16 weeks will include exercise programmes of 48 sessions conducted three times per week for two of the three study groups. These groups will be: a group participating in a conventional training programme, based on a preplanned intensity progression; and, a group of participants involved in an exercise programme which will vary the exercise intensity regarding patients' daily Heart Rate Variability. Each session will include a warm-up, the main part of cardiovascular and strength training and a cool-down including stretching exercises.

All the participants will be evaluated before and after the intervention measuring clinical, physical and psychosocial assessments. The clinical variables will be evaluated in patients' reference hospital and will involve medical history registers, cardiotoxicity variables, blood analysis and inflammatory factors measures. Physical and psychosocial variables measurement will be carried out in a sports centre and will include the assessment of: body composition, heart rate variability, cardiorespiratory capacity, upper and lower extremities' strength and flexibility, agility and balance, quality of life, fatigue, functionality, life satisfaction, self-esteem, anxiety and depression, shoulder mobility perception, kinesiophobia, physical activity level and exercise motivation.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 65 years
* Being a breast cancer patient with luminal or triple-negative
* Having completed the radiotherapy treatment, after chemotherapy, approximately one month ago.
* Be able to perform the proposed tests safely

Exclusion Criteria:

* Being undergoing radiotherapy treatment or scheduled for surgery
* Having metastasic cancer
* Not having any serious psychiatric illness

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-09-13 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
Baseline Troponin | At baseline
  A haemogram will be carried out to analyse patients' Troponin I and T to detect their cardiotoxicity levels. Troponin results will be reported in ng/L.
After intervention Troponin | Immediately after the intervention
  A haemogram will be carried out to analyse patients' Troponin I and T to detect their cardiotoxicity levels and the change produced after the intervention. Troponin results will be reported in ng/L.
3 months after intervention Troponin | 3 months after the intervention ending
  A haemogram will be carried out to analyse patients' Troponin I and T to detect their cardiotoxicity levels and the changes produced 3 months after the intervention. Troponin results will be reported in ng/L.
6 months after intervention Troponin | 6 months after the intervention ending
  A haemogram will be carried out to analyse patients' Troponin I and T to detect their cardiotoxicity levels and the changes produced 6 months after the intervention. Troponin results will be reported in ng/L.
Baseline Brain Natriuretic Peptide | At baseline
  A haemogram will be carried out to analyse patients' BNP to assess their cardiotoxicity levels. BNP results will be reported in pg/ml.
After intervention Brain Natriuretic Peptide | Immediately after the intervention
  A haemogram will be carried out to analyse patients' BNP to assess their cardiotoxicity levels and the change produced after the intervention. BNP results will be reported in pg/ml.
3 months after intervention Brain Natriuretic Peptide | 3 months after the intervention ending
  A haemogram will be carried out to analyse patients' BNP to assess their cardiotoxicity levels and the change produced 3 after the intervention. BNP results will be reported in pg/ml.
6 months after intervention Brain Natriuretic Peptide | 6 months after the intervention ending
  A haemogram will be carried out to analyse patients' BNP to assess their cardiotoxicity levels and the change produced 6 after the intervention. BNP results will be reported in pg/ml.
Baseline left ventricular systolic and diastolic volume | At Baseline
  An echocardiogram will be performed to measure left ventricular systolic and diastolic volume in mL.
After intervention left ventricular systolic and diastolic volume | Immediately after the intervention ending
  An echocardiogram will be performed to measure left ventricular systolic and diastolic volume in mL and it changes after the intervention.
3 months after intervention left ventricular systolic and diastolic volume | 3 months after the intervention ending
  An echocardiogram will be performed to measure left ventricular systolic and diastolic volume in mL and it changes 3 months after the intervention.
6 months after intervention left ventricular systolic and diastolic volume | 6 months after the intervention ending
  An echocardiogram will be performed to measure left ventricular systolic and diastolic volume in mL and it changes 6 months after the intervention.
Baseline left ventricular ejection fraction | At baseline
  By an echocardiogram, patients' % of LVEF will be assessed due to its possible modification caused by cardiotoxicity.
After intervention left ventricular ejection fraction | Immediately after the intervention
  By an echocardiogram, patients' % of LVEF will be assessed to measure its results and its change after the intervention.
3 months after intervention left ventricular ejection fraction | 3 months after the intervention ending
  By an echocardiogram, patients' % of LVEF will be assessed to measure its results and its change 3 months after the intervention.
6 months after intervention left ventricular ejection fraction | 6 months after the intervention ending
  By an echocardiogram, patients' % of LVEF will be assessed to measure its results and its change 6 months after the intervention.
Baseline time domain heart rate variability measures | At baseline
  The assessment of heart rate variability will be performed with a Polar chest strap and electrocardiogram. Participants will remain in the supine position for 10 minutes to correctly obtain 5 minutes of a stable signal. After removal of artefacts, the standard deviation time domains of all RR intervals (SDNN) in ms, the mean ad all RR intervals in ms and the root mean square of the sum of squared RR interval differences in ms (RMSSD) will be recorded.
After intervention time-domain heart rate variability measures | Immediately after the intervention
  The assessment of heart rate variability will be performed with a Polar chest strap and electrocardiogram. Participants will remain in the supine position for 10 minutes to correctly obtain 5 minutes of a stable signal. After removal of artefacts, the standard deviation time domains of all RR intervals (SDNN) in ms, the mean ad all RR intervals in ms and the root mean square of the sum of squared RR interval differences in ms (RMSSD) will be recorded after the intervention.
3 months after intervention time-domain heart rate variability measures | 3 months after the intervention ending
  The assessment of heart rate variability will be performed with a Polar chest strap and electrocardiogram. Participants will remain in the supine position for 10 minutes to correctly obtain 5 minutes of a stable signal. After removal of artefacts, the standard deviation time domains of all RR intervals (SDNN) in ms, the mean ad all RR intervals in ms and the root mean square of the sum of squared RR interval differences in ms (RMSSD) will be recorded 3 months after the intervention.
6 months after intervention time-domain heart rate variability measures | 6 months after the intervention ending
  The assessment of heart rate variability will be performed with a Polar chest strap and electrocardiogram. Participants will remain in the supine position for 10 minutes to correctly obtain 5 minutes of a stable signal. After removal of artefacts, the standard deviation time domains of all RR intervals (SDNN) in ms, the mean ad all RR intervals in ms and the root mean square of the sum of squared RR interval differences in ms (RMSSD) will be recorded 6 months after the intervention.
During intervention time-domain heart rate variability measures | During the intervention ending
  Daily heart rate variability will be measured using the HRV4Training application, a validated mobile application that allows HRV values to be obtained by photoplethysmography (rMSSD, SDNN, AVNN, pNN50 and heart rate).
Baseline frequency domain heart rate variability measures | At baseline
  The assessment of heart rate variability will be performed with a Polar chest strap and electrocardiogram. Participants will remain in the supine position for 10 minutes to correctly obtain 5 minutes of a stable signal. After removal of artefacts, the frequency measures of low frequency (LF, 0.04-0.15 Hz) in ms2 and n.u, high frequency (HF, 0.15-0.4 Hz) ms2 and n.u, total power in ms2 and LF/HF ratio will be calculated.
After intervention frequency domain heart rate variability measures | Immediately after the intervention
  The assessment of heart rate variability will be performed with a Polar chest strap and electrocardiogram. Participants will remain in the supine position for 10 minutes to correctly obtain 5 minutes of a stable signal. After removal of artefacts, the frequency measures of low frequency (LF, 0.04-0.15 Hz) in ms2 and n.u, high frequency (HF, 0.15-0.4 Hz) ms2 and n.u, total power in ms2 and LF/HF ratio will be calculated after intervention.
3 months after intervention frequency domain heart rate variability measures | 3 months after the intervention ending
  The assessment of heart rate variability will be performed with a Polar chest strap and electrocardiogram. Participants will remain in the supine position for 10 minutes to correctly obtain 5 minutes of a stable signal. After removal of artefacts, the frequency measures of low frequency (LF, 0.04-0.15 Hz) in ms2 and n.u, high frequency (HF, 0.15-0.4 Hz) ms2 and n.u, total power in ms2 and LF/HF ratio will be calculated 3 months after the intervention.
6 months after intervention frequency domain heart rate variability measures | 6 months after the intervention ending
  The assessment of heart rate variability will be performed with a Polar chest strap and electrocardiogram. Participants will remain in the supine position for 10 minutes to correctly obtain 5 minutes of a stable signal. After removal of artefacts, the frequency measures of low frequency (LF, 0.04-0.15 Hz) in ms2 and n.u, high frequency (HF, 0.15-0.4 Hz) ms2 and n.u, total power in ms2 and LF/HF ratio will be calculated 6 months after the intervention.
During intervention frequency domain heart rate variability measures | During the intervention
  Daily heart rate variability will be measured using the HRV4Training application, a validated mobile application that allows HRV values to be obtained by photoplethysmography (LF, HF, TP, LF/HF and recovery points)

SECONDARY OUTCOMES:
Baseline heart rate rhyme | At baseline
  A resting electrocardiogram will be used to obtain patients' normal values for heart rate measurements in bpm, I-axis and aVF, Q-T interval, QRS complex, S-T segment and T-wave, in ms. Moreover, resting heart rate will be assessed by a Polar chest band.
After intervention heart rate rhyme | Immediately after the intervention
  A resting electrocardiogram will be used to obtain patients' normal values for heart rate measurements in bpm, I-axis and aVF, Q-T interval, QRS complex, S-T segment and T-wave, in ms, and get after intervention results. Moreover, resting heart rate will be assessed by a Polar chest band.
3 months after intervention heart rate rhyme | 3 months after the intervention ending
  A resting electrocardiogram will be used to obtain patients' normal values for heart rate measurements in bpm, I-axis and aVF, Q-T interval, QRS complex, S-T segment and T-wave, in ms, and get its results 3 months after the intervention. Moreover, resting heart rate will be assessed by a Polar chest band.
6 months after intervention heart rate rhyme | 6 months after the intervention
  A resting electrocardiogram will be used to obtain patients' normal values for heart rate measurements in bpm, I-axis and aVF, Q-T interval, QRS complex, S-T segment and T-wave, in ms, and get its results 6 months after the intervention. Moreover, resting heart rate will be assessed by a Polar chest band.
Baseline tumor necrosis factor | At baseline
  Through a blood analysis TFN, in pg/mL, will be measured to evaluate patients' inflammation.
After intervention tumor necrosis factor | Immediately after the intervention
  Through a blood analysis TFN, in pg/mL, will be measured to evaluate patients' inflammation after the intervention.
3 months after intervention tumor necrosis factor | 3 months after the intervention ending
  Through a blood analysis TFN, in pg/mL, will be measured to evaluate patients' inflammation 3 months after the intervention.
6 months after intervention tumor necrosis factor | 6 months after the intervention ending
  Through a blood analysis TFN, in pg/mL, will be measured to evaluate patients' inflammation 6 months after the intervention.
Baseline interleukins measurement | At baseline
  The inflammation will be assessed by blood interleukins will include IL-6, IL-8, IL-1b, IL-1ra and IL-10 values, in pg/m.
After intervention interleukins measurement | Immediately after the intervention.
  The inflammation will be assessed by blood interleukins will include IL-6, IL-8, IL-1b, IL-1ra and IL-10 values, in pg/m, immediately after the intervention.
3 months after intervention interleukins measurement | 3 months after the intervention ending
  The inflammation will be assessed by blood interleukins will include IL-6, IL-8, IL-1b, IL-1 and IL-10 values, in pg/m, 3 months after the intervention.
6 months after intervention interleukins measurement | 6 months after the intervention ending
  The inflammation will be assessed by blood interleukins will include IL-6, IL-8, IL-1b, IL-1ra and IL-10 values, in pg/m, 6 months after the intervention.
Baseline C-reactive protein measure | At baseline
  C-reactive protein (CRP), measured in mg/L will be evaluated to get patients' pro-inflammatory data.
After intervention C-reactive protein measure | Immediately after the intervention.
  C-reactive protein (CRP), measured in mg/L will be evaluated to get patients' pro-inflammatory data after the intervention.
3 months after intervention C-reactive protein measure | 3 months after the intervention ending
  C-reactive protein (CRP), measured in mg/L will be evaluated to get patients' pro-inflammatory data 3 months after the intervention.
6 months after intervention C-reactive protein measure | 6 months after the intervention ending
  C-reactive protein (CRP), measured in mg/L will be evaluated to get patients' pro-inflammatory data 6 months after the intervention.
Baseline monocyte chemotactic protein measure | At baseline
  Monocyte chemotactic protein (MCP-1), measured in pg/mL will be evaluated to get patients' pro-inflammatory data.
After intervention monocyte chemotactic protein measure | Immediately after the intervention.
  Monocyte chemotactic protein (MCP-1), measured in pg/mL will be evaluated to get patients' pro-inflammatory data after the intervention.
3 months after intervention monocyte chemotactic protein measure | 3 months after the intervention ending
  Monocyte chemotactic protein (MCP-1), measured in pg/mL will be evaluated to get patients pro-inflammatory data 3 months after the intervention.
6 months after intervention monocyte chemotactic protein measure | 6 months after the intervention ending
  Monocyte chemotactic protein (MCP-1), measured in pg/mL will be evaluated to get patients pro-inflammatory data 6 months after the intervention.
Baseline glucose measure | At baseline
  Glucose, in mg/dl, will be measure through a blood test due to be related to cancer prognosis and cardiovascular risk.
After intervention glucose measure | Immediately after the intervention.
  Glucose, in mg/dl, will be measure after intervention through a blood test due to be related to cancer prognosis and cardiovascular risk.
3 months after intervention glucose measure | 3 months after the intervention ending
  Glucose, in mg/dl, will be measure through a blood test due to be related to cancer prognosis and cardiovascular risk.
6 months after intervention glucose measure | 6 months after the intervention ending
  Glucose, in mg/dl, will be measure through a blood test due to be related to cancer prognosis and cardiovascular risk.
Baseline cholesterol measure | At baseline
  Low-density lipoprotein and high-density lipoprotein, measured in mg/dL, will be assessed by a blood test due to be related to cancer prognosis and cardiovascular risk.
After intervention cholesterol measure | Immediately after the intervention.
  Low-density lipoprotein and high-density lipoprotein, measured in mg/dL, will be measure after intervention by a blood test due to be related to cancer prognosis and cardiovascular risk.
3 months after intervention cholesterol measure | 3 months after the intervention ending
  Low-density lipoprotein and high-density, measured in mg/dL, will be measure 3 months after the intervention by a blood test due to be related to cancer prognosis and cardiovascular risk.
6 months after intervention cholesterol measure | 6 months after the intervention ending
  Low-density lipoprotein and high-density, measured in mg/dL, will be measure 6 months after the intervention by a blood test due to be related to cancer prognosis and cardiovascular risk.
Baseline blood pressure measures | At baseline
  Measurements of blood pressure will be performed using a validated oscillometer. Participants will remain at rest for five minutes before the assessment. They will place their left arm, on which the measurement will be taken, on the table so that the cuff is at the level of the heart, 2 cm from the elbow. In addition, any clothing that may alter the results shall be removed. Once in this position, the air tube of the cuff shall be placed on the front of the upper arm in line with the middle finger and the blue arrow on the cuff. Systolic and diastolic blood pressure data, measured in mmHg, shall be taken, and then the mean arterial pressure = (systolic blood pressure+ (2*diastolic blood pressure))/3 shall be calculated.
After intervention blood pressure measures | Immediately after the intervention.
  Measurements of blood pressure after the intervention will be performed using a validated oscillometer. Participants will remain at rest for five minutes before the assessment. They will place their left arm, on which the measurement will be taken, on the table so that the cuff is at the level of the heart, 2 cm from the elbow. In addition, any clothing that may alter the results shall be removed. Once in this position, the air tube of the cuff shall be placed on the front of the upper arm in line with the middle finger and the blue arrow on the cuff. Systolic and diastolic blood pressure data, measured in mmHg, shall be taken, and then the mean arterial pressure = (systolic blood pressure+ (2*diastolic blood pressure))/3 shall be calculated.
3 months after intervention blood pressure measures | 3 months after the intervention ending
  Measurements of blood pressure 3 months after the intervention will be performed using a validated oscillometer. Participants will remain at rest for five minutes before the assessment. They will place their left arm, on which the measurement will be taken, on the table so that the cuff is at the level of the heart, 2 cm from the elbow. In addition, any clothing that may alter the results shall be removed. Once in this position, the air tube of the cuff shall be placed on the front of the upper arm in line with the middle finger and the blue arrow on the cuff. Systolic and diastolic blood pressure data, measured in mmHg, shall be taken, and then the mean arterial pressure = (systolic blood pressure+ (2*diastolic blood pressure))/3 shall be calculated.
6 months after intervention blood pressure measures | 6 months after the intervention ending
  Measurements of blood pressure 6 months after the intervention will be performed using a validated oscillometer. Participants will remain at rest for five minutes before the assessment. They will place their left arm, on which the measurement will be taken, on the table so that the cuff is at the level of the heart, 2 cm from the elbow. In addition, any clothing that may alter the results shall be removed. Once in this position, the air tube of the cuff shall be placed on the front of the upper arm in line with the middle finger and the blue arrow on the cuff. Systolic and diastolic blood pressure data, measured in mmHg, shall be taken, and then the mean arterial pressure = (systolic blood pressure+ (2*diastolic blood pressure))/3 shall be calculated.
Baseline body composition weight measures | At baseline
  The weight assessment of body composition will be performed by impedance to obtain patients' global bodyweight, musculoskeletal mass, mineral mass, fat mass and upper and lower extremities segmental fat and lean mass weight. All the measures will be reported in kilograms.
After intervention body composition weight measures | Immediately after the intervention.
  The weight assessment of body composition after the intervention will be performed by impedance to obtain patients' global bodyweight, musculoskeletal mass, mineral mass, fat mass and upper and lower extremities segmental fat and lean mass weight. All the measures will be reported in kilograms.
3 months after intervention body composition weight measures | 3 months after the intervention ending
  The weight assessment of body composition 3 months after the intervention will be performed by impedance to obtain patients' global bodyweight, musculoskeletal mass, mineral mass, fat mass and upper and lower extremities segmental fat and lean mass weight. All the measures will be reported in kilograms.
6 months after intervention body composition weight measures | 6 months after the intervention ending
  The weight assessment of body composition 6 months after the intervention will be performed by impedance to obtain patients' global bodyweight, musculoskeletal mass, mineral mass, fat mass and upper and lower extremities segmental fat and lean mass weight. All the measures will be reported in kilograms
Baseline body composition percentages measures | At baseline
  The assessment of the body fat percentage of the participants is a variable to be taken into consideration. Therefore, thought impedance patients' body fat percentage and upper and lower extremities segmental fat and lean mass percentages will be recorded.
After intervention body composition percentages measures | Immediately after the intervention.
  The assessment of the body percentage of the participants is a variable to be taken into consideration. Therefore, thought impedance, patients' body fat percentage and upper and lower extremities segmental fat and lean mass percentages will be recorded after the intervention.
3 months after intervention body composition percentages measures | 3 months after the intervention ending
  The assessment of the body percentage of the participants is a variable to be taken into consideration. Therefore, thought impedance, patients' body fat percentage and upper and lower extremities segmental fat and lean mass percentages will be recorded 3 months after the intervention.
6 months after intervention body composition percentages measures | 6 months after the intervention ending
  The assessment of the body percentage of the participants is a variable to be taken into consideration. Therefore, thought impedance, patients' body fat percentage and upper and lower extremities segmental fat and lean mass percentages will be recorded 6 months after the intervention.
Baseline body water measures | At baseline
  By employing also impedance body water evaluation, measured in liters, will be carried out.
After intervention body water measures | Immediately after the intervention.
  By employing also impedance, body water evaluation, measured in liters, will be carried out after the intervention.
3 months after intervention body water measures | 3 months after the intervention ending
  By employing also impedance, body water evaluation, measured in liters, will be carried out 3 months after the intervention.
6 months after intervention body water measures | 6 months after the intervention ending
  By employing also impedance, body water evaluation, measured in liters, will be carried out 6 months after the intervention.
Baseline anthropometric measures | At baseline
  Patients' height and body perimeters will be assessed in centimeters. Especially, waist circumference, hip circumference, arm circumferences, leg circumferences will be measured following the guidelines set by the American College of Sports Medicine. Afterward, patients' height will be used together with their corresponding weight to calculate patients Body Mass Index.
After intervention anthropometric measures | Immediately after the intervention.
  Patients' height and body perimeters will be assessed in centimeters immediately after the intervention. Especially, waist circumference, hip circumference, arm circumferences, leg circumferences will be measured following the guidelines set by the American College of Sports Medicine. Afterward, patients' height will be used together with their corresponding weight to calculate patients Body Mass Index.
3 months after intervention anthropometric measures | 3 months after the intervention ending
  Patients' height and body perimeters will be assessed in centimeters 3 months after the end of the intervention. Especially, waist circumference, hip circumference, arm circumferences, leg circumferences will be measured following the guidelines set by the American College of Sports Medicine. Afterward, patients' height will be used together with their corresponding weight to calculate patients Body Mass Index.
6 months after intervention anthropometric measures | 6 months after the intervention ending
  Patients' height and body perimeters will be assessed in centimeters 6 months after the end of the intervention. Especially, waist circumference, hip circumference, arm circumferences, leg circumferences will be measured following the guidelines set by the American College of Sports Medicine. Afterward, patients' height will be used together with their corresponding weight to calculate patients Body Mass Index.
Baseline cardiorespiratory fitness | At baseline
  To record cardiorespiratory fitness, maximum heart rate and patients' perception of exertion, the Bruce incremental submaximal test (modified) was performed on a treadmill. During the test, the patients will wear a chest strap for heart rate monitoring. Thus, following the protocol created by Bruce, the treadmill will start with a 0% incline and a speed of 1.7 m/h which will be maintained for the first 3 minutes. Every 3 minutes, both the speed and the incline will be increased until the participants decide that their fatigue is too great to continue. At the end of the test, the recovery heart rate is recorded 1 minute after stopping the test to assess the recovery rate. Subsequently, the maximum oxygen consumption of each patient (VO2max = 2.282* (time) + 8.545) will be calculated from the formula proposed by the creators.
After intervention cardiorespiratory fitness | Immediately after the intervention.
  To record cardiorespiratory fitness after the intervention, maximum heart rate and patients' perception of exertion, the Bruce incremental submaximal test (modified) was performed on a treadmill. During the test, the patients will wear a chest strap for heart rate monitoring. Thus, following the protocol created by Bruce, the treadmill will start with a 0% incline and a speed of 1.7 m/h which will be maintained for the first 3 minutes. Every 3 minutes, both the speed and the incline will be increased until the participants decide that their fatigue is too great to continue. At the end of the test, the recovery heart rate is recorded 1 minute after stopping the test to assess the recovery rate. Subsequently, the maximum oxygen consumption of each patient (VO2max = 2.282* (time) + 8.545) will be calculated from the formula proposed by the creators.
3 months after intervention cardiorespiratory fitness | 3 months after the intervention ending
  To record cardiorespiratory fitness 3 months after the intervention, maximum heart rate and patients' perception of exertion, the Bruce incremental submaximal test (modified) was performed on a treadmill. During the test, the patients will wear a chest strap for heart rate monitoring. Thus, following the protocol created by Bruce, the treadmill will start with a 0% incline and a speed of 1.7 m/h which will be maintained for the first 3 minutes. Every 3 minutes, both the speed and the incline will be increased until the participants decide that their fatigue is too great to continue. At the end of the test, the recovery heart rate is recorded 1 minute after stopping the test to assess the recovery rate. Subsequently, the maximum oxygen consumption of each patient (VO2max = 2.282* (time) + 8.545) will be calculated from the formula proposed by the creators.
6 months after intervention cardiorespiratory fitness | 6 months after the intervention ending
  To record cardiorespiratory fitness 6 months after the intervention, maximum heart rate and patients' perception of exertion, the Bruce incremental submaximal test (modified) was performed on a treadmill. During the test, the patients will wear a chest strap for heart rate monitoring. Thus, following the protocol created by Bruce, the treadmill will start with a 0% incline and a speed of 1.7 m/h which will be maintained for the first 3 minutes. Every 3 minutes, both the speed and the incline will be increased until the participants decide that their fatigue is too great to continue. At the end of the test, the recovery heart rate is recorded 1 minute after stopping the test to assess the recovery rate. Subsequently, the maximum oxygen consumption of each patient (VO2max = 2.282* (time) + 8.545) will be calculated from the formula proposed by the creators.
Baseline measurement of lower-body strength endurance | At baseline
  Functional strength will be measure by the 30 seconds chair stand test. The patient will stand up, position herself fully stretched, and perform as many repetitions as possible in 30 seconds.
After intervention measurement of lower-body strength endurance | Immediately after the intervention.
  Functional strength will be measure by the 30 seconds chair stand test. The patient will stand up, position herself fully stretched, and perform as many repetitions as possible in 30 seconds.
3 months after intervention measurement of lower-body strength endurance | 3 months after the intervention ending
  Functional strength will be measure by the 30 seconds chair stand test. The patient will stand up, position herself fully stretched, and perform as many repetitions as possible in 30 seconds.
6 months after intervention measurement of lower-body strength endurance | 6 months after the intervention ending
  Functional strength will be measure by the 30 seconds chair stand test. The patient will stand up, positioning herself fully stretched, and perform as many repetitions as possible in 30 seconds.
Baseline maximal strength | At baseline
  The evaluation of maximal strength will be performed by using an encoder for the correct calculation of the Maximum Repetition (RM) from the speed and power generated by moving the weight vertically. The participants will perform 4 tests to assess the different muscular groups' strength (Back Squat Test, Deadlift Test, Lunge Test, Barbell Hip Thrust Test). Concretely, 4-5 repetitions will be performed with incremental weights where the speed of execution decreases.
After intervention maximal strength | Immediately after the intervention.
  The evaluation of maximal strength after the intervention will be performed by using an encoder for the correct calculation of the Maximum Repetition (RM) from the speed and power generated by moving the weight vertically. The participants will perform 4 tests to assess the different muscular groups' strength (Back Squat Test, Deadlift Test, Lunge Test, Barbell Hip Thrust Test). Concretely, 4-5 repetitions will be performed with incremental weights where the speed of execution decreases.
3 months after intervention maximal strength | 3 months after the intervention ending
  The evaluation of maximal strength 3 months after the intervention will be performed by using an encoder for the correct calculation of the Maximum Repetition (RM) from the speed and power generated by moving the weight vertically. The participants will perform 4 tests to assess the different muscular groups' strength (Back Squat Test, Deadlift Test, Lunge Test, Barbell Hip Thrust Test). Concretely, 4-5 repetitions will be performed with incremental weights where the speed of execution decreases.
6 months after intervention maximal strength | 6 months after the intervention ending
  The evaluation of maximal strength 6 months after the intervention will be performed by using an encoder for the correct calculation of the Maximum Repetition (RM) from the speed and power generated by moving the weight vertically. The participants will perform 4 tests to assess the different muscular groups' strength (Back Squat Test, Deadlift Test, Lunge Test, Barbell Hip Thrust Test). Concretely, 4-5 repetitions will be performed with incremental weights where the speed of execution decreases.
Baseline vertical applied force | At baseline
  The force-power will be measured using a countermovement jump test (CMJ) and squat jump test (SJ). From these tests, the maximum force (N) and power (P) exerted during impulse and landing, flight time (ms) and jump height (cm) will be obtained. For the evaluation of the different variables indicated, different technologies will be used such as a jump platform and/or the recording of each of the jumps for subsequent analysis with the validated application of My Jump and Kinovea.
After intervention vertical applied force | Immediately after the intervention.
  The after-intervention force-power will be measured using a countermovement jump test (CMJ) and squat jump test (SJ). From these tests, the maximum force (N) and power (P) exerted during impulse and landing, flight time (ms) and jump height (cm) will be obtained. For the evaluation of the different variables indicated, different technologies will be used such as a jump platform and/or the recording of each of the jumps for subsequent analysis with the validated application of My Jump and Kinovea.
3 months intervention vertical applied force | 3 months after the intervention ending
  The force-power 3 months after the intervention will be measured using a countermovement jump test (CMJ) and squat jump test (SJ). From these tests, the maximum force (N) and power (P) exerted during impulse and landing, flight time (ms) and jump height (cm) will be obtained. For the evaluation of the different variables indicated, different technologies will be used such as a jump platform and/or the recording of each of the jumps for subsequent analysis with the validated application of My Jump and Kinovea.
6 months intervention vertical applied force | 6 months after the intervention ending
  The force-power 6 months after the intervention will be measured using a countermovement jump test (CMJ) and squat jump test (SJ). From these tests, the maximum force (N) and power (P) exerted during impulse and landing, flight time (ms) and jump height (cm) will be obtained. For the evaluation of the different variables indicated, different technologies will be used such as a jump platform and/or the recording of each of the jumps for subsequent analysis with the validated application of My Jump and Kinovea.
Baseline measurement of upper body strength endurance | At baseline
  The strength endurance of the patients will be measured utilizing the 30-second arm curl test reporting the maximum number of repetitions in 30 seconds.
After intervention measurement of upper body strength endurance | Immediately after the intervention.
  The strength endurance of the patients after the intervention will be measured employing the 30-second arm curl test reporting the maximum number of repetitions in 30 seconds.
3 months after intervention measurement of upper body strength endurance | 3 months after the intervention ending
  The strength endurance of the patients 3 months after the intervention will be measured utilizing the 30-second arm curl test reporting the maximum number of repetitions in 30 seconds.
6 months after intervention measurement of upper body strength endurance | 6 months after the intervention ending
  The strength endurance of the patients 6 months after the intervention will be measured employing the 30-second arm curl test reporting the maximum number of repetitions in 30 seconds.
Baseline maximal upper body strength | At baseline
  Maximal strength of different muscular group exercises will be assessed (chest press, shoulder press, bent over row, biceps curl with barbell, Triceps extension with barbell) based on the number of repetitions that the participants are able to perform. An encoder will be used to calculate the Maximum Repetition (RM) by the speed and power generated by moving the weight vertically.
After intervention maximal upper body strength | Immediately after the intervention.
  Maximal strength of different muscular group exercises after the intervention will be assessed (chest press, shoulder press, bent over row, biceps curl with barbell, Triceps extension with barbell) based on the number of repetitions that the participants are able to perform. An encoder will be used to calculate the Maximum Repetition (RM) by the speed and power generated by moving the weight vertically.
3 months after intervention maximal upper body strength | 3 months after the intervention ending
  Maximal strength of different muscular group exercises 3 months after the intervention will be assessed (chest press, shoulder press, bent over row, biceps curl with barbell, Triceps extension with barbell) based on the number of repetitions that the participants are able to perform. An encoder will be used to calculate the Maximum Repetition (RM) by the speed and power generated by moving the weight vertically.
6 months after intervention maximal upper body strength | 6 months after the intervention ending
  Maximal strength of different muscular group exercises 6 months after the intervention will be assessed (chest press, shoulder press, bent over row, biceps curl with barbell, Triceps extension with barbell) based on the number of repetitions that the participants are able to perform. An encoder will be used to calculate the Maximum Repetition (RM) by the speed and power generated by moving the weight vertically.
Baseline measurement of agility and dynamic balance | At baseline
  The 8-foot up-and-go test will be employed to measure dynamic balance and agility, where the participants will get up from the chair and walk as fast as possible to the cone, placed 2,44 meters far away, and around the cone, back to the chair. The outcome measure will be the time spend in seconds.
After intervention measurement of agility and dynamic balance | Immediately after the intervention.
  The 8-foot up-and-go test will be employed to measure dynamic balance and agility after the intervention, where the participants will get up from the chair and walk as fast as possible to the cone, placed 2,44 meters far away, and around the cone, back to the chair. The outcome measure will be the time spend in seconds.
3 months after intervention measurement of agility and dynamic balance | 3 months after the intervention ending
  The 8-foot up-and-go test will be employed to measure dynamic balance and agility 3 months after the intervention, where the participants will get up from the chair and walk as fast as possible to the cone, placed 2,44 meters far away, and around the cone, back to the chair. The outcome measure will be the time spend in seconds.
6 months after intervention measurement of agility and dynamic balance | 6 months after the intervention ending
  The 8-foot up-and-go test will be employed to measure dynamic balance and agility 6 months after the intervention, where the participants will get up from the chair and walk as fast as possible to the cone, placed 2,44 meters far away, and around the cone, back to the chair. The outcome measure will be the time spend in seconds.
Baseline static monopodal balance | At baseline
  The one-leg stand test from the adults ALHPA battery will assess static balance. For this purpose, the patient will be placed in monopodal support, placing the sole on the inside of the knee. The time reached, in seconds, without touching the group with the other foot will be recorded.
After intervention static monopodal balance | Immediately after the intervention.
  The one-leg stand test from the adults ALHPA battery will assess static balance after the intervention. For this purpose, the patient will be placed in monopodal support, placing the sole of the foot on the inside of the knee. The time reached, in seconds, without touching the group with the other foot will be recorded.
3 months after intervention static monopodal balance | 3 months after the intervention ending
  The one-leg stand test from the adults ALHPA battery will assess static balance 3 months after the intervention. For this purpose, the patient will be placed in monopodal support, placing the sole on the inside of the knee. The time reached, in seconds, without touching the group with the other foot will be recorded.
6 months after intervention static monopodal balance | 6 months after the intervention ending
  The one-leg stand test from the adults ALHPA battery will assess static balance 6 months after the intervention. For this purpose, the patient will be placed in monopodal support, placing the sole of the foot on the inside of the knee. The time reached, in seconds, without touching the group with the other foot will be recorded
Baseline measurement of upper body flexibility | At baseline
  Flexibility will be assessed using the Back scratch test, previously used in breast cancer patients and belonging to the Senior Fitness Test battery. During the test, participants will stand upright and try to reach over their head, with their arm in flexion and external rotation, to touch their other hand, which will be placed on their back in a supine position with the arm flexed. The centimeters left or passed from one hand to the other will be noted.
After intervention measurement of upper body flexibility | Immediately after the intervention.
  Flexibility after the intervention will be assessed using the Back scratch test, previously used in breast cancer patients and belonging to the Senior Fitness Test battery. During the test, participants will stand upright and try to reach over their head, with their arm in flexion and external rotation, to touch their other hand, which will be placed on their back in a supine position with the arm flexed. The centimeters left or passed from one hand to the other will be noted.
3 months after intervention measurement of upper body flexibility | 3 months after the intervention ending
  Flexibility 3 months after the intervention will be assessed using the Back scratch test, previously used in breast cancer patients and belonging to the Senior Fitness Test battery. During the test, participants will stand upright and try to reach over their head, with their arm in flexion and external rotation, to touch their other hand, which will be placed on their back in a supine position with the arm flexed. The centimeters left or passed from one hand to the other will be noted.
6 months after intervention measurement of upper body flexibility | 6 months after the intervention ending
  Flexibility 6 months after the intervention will be assessed using the Back scratch test, previously used in breast cancer patients and belonging to the Senior Fitness Test battery. During the test, participants will stand upright and try to reach over their head, with their arm in flexion and external rotation, to touch their other hand, which will be placed on their back in a supine position with the arm flexed. The centimeters left or passed from one hand to the other will be noted.
Baseline measurement of lower body flexibility | At baseline
  Hamstring flexibility will be measured using the V Sit and Reach test where the participant will be seated on the floor with knees fully extended and feet 30 cm apart. A tape measure will be placed on the floor, equidistant between the feet, placing the 0 cm in line with the heels. Pressing the palms of the hands together and keeping the elbows fully extended, the participants shall bend their trunk as far as possible over the tape measure. The results will be expressed in centimeters reporting the distance left or passed from the feet.
After intervention measurement of lower body flexibility | Immediately after the intervention.
  Hamstring flexibility after the intervention will be measured using the V Sit and Reach test where the participant will be seated on the floor with knees fully extended and feet 30 cm apart. A tape measure will be placed on the floor, equidistant between the feet, placing the 0 cm in line with the heels. Pressing the palms of the hands together and keeping the elbows fully extended, the participants shall bend their trunk as far as possible over the tape measure. The results will be expressed in centimeters reporting the distance left or passed from the feet.
3 months after intervention measurement of lower body flexibility | 3 months after the intervention ending
  Hamstring flexibility 3 months after the intervention will be measured using the V Sit and Reach test where the participant will be seated on the floor with knees fully extended and feet 30 cm apart. A tape measure will be placed on the floor, equidistant between the feet, placing the 0 cm in line with the heels. Pressing the palms of the hands together and keeping the elbows fully extended, the participants shall bend their trunk as far as possible over the tape measure. The results will be expressed in centimeters reporting the distance left or passed from the feet.
6 months after intervention measurement of lower body flexibility | 6 months after the intervention ending
  Hamstring flexibility 6 months after the intervention will be measured using the V Sit and Reach test where the participant will be seated on the floor with knees fully extended and feet 30 cm apart. A tape measure will be placed on the floor, equidistant between the feet, placing the 0 cm in line with the heels. Pressing the palms of the hands together and keeping the elbows fully extended, the participants shall bend their trunk as far as possible over the tape measure. The results will be expressed in centimeters reporting the distance left or passed from the feet.
Baseline health-related quality of life measure | At baseline
  Psychological variables will be assessed employing self-administered questionnaires specifically validated for cancer patients. Health-related quality of life will be assessed using the EORTC QLQ-C30 Quality of Life Questionnaire which includes functional and cancer-specific symptom assessment. Higher global scores will mean a higher quality of life.
After intervention health-related quality of life measure | Immediately after the intervention.
  Psychological variables will be assessed employing self-administered questionnaires specifically validated for cancer patients. Health-related quality of life will be assessed using the EORTC QLQ-C30 Quality of Life Questionnaire which includes functional and cancer-specific symptom assessment. Higher global scores will mean a higher quality of life.
3 months after intervention health-related quality of life measure | 3 months after the intervention ending
  Psychological variables will be assessed utilizing self-administered questionnaires specifically validated for cancer patients. Health-related quality of life will be assessed 3 months after the intervention using the EORTC QLQ-C30 Quality of Life Questionnaire which includes functional and cancer-specific symptom assessment. Higher global scores will mean a higher quality of life.
6 months after intervention health-related quality of life measure | 6 months after the intervention ending
  Psychological variables will be assessed through self-administered questionnaires specifically validated for cancer patients. Health-related quality of life 6 months after the intervention will be assessed using the EORTC QLQ-C30 Quality of Life Questionnaire which includes functional and cancer-specific symptom assessment. Higher global scores will mean a higher quality of life.
Baseline cancer-related fatigue | At baseline
  To assess cancer-related fatigue, the FACT-F questionnaire will be employed. It includes 13 items where patients will select their fatigue perception with a Likert scale from 1 to 5 being 1 the lowest fatigue score and 5 the highest.
After intervention cancer-related fatigue | Immediately after the intervention.
  To assess cancer-related fatigue after the intervention, the FACT-F questionnaire will be employed. It includes 13 items where patients will select their fatigue perception with a Likert scale from 1 to 5 being 1 the lowest fatigue score and 5 the highest.
3 months after intervention cancer-related fatigue | 3 months after the intervention ending
  To assess cancer-related fatigue 3 months after the intervention, the FACT-F questionnaire will be employed. It includes 13 items where patients will select their fatigue perception with a Likert scale from 1 to 5 being 1 the lowest fatigue score and 5 the highest.
6 months after intervention cancer-related fatigue | 6 months after the intervention ending
  To assess cancer-related fatigue 6 months after the intervention, the FACT-F questionnaire will be employed. It includes 13 items where patients will select their fatigue perception with a Likert scale from 1 to 5 being 1 the lowest fatigue score and 5 the highest.
Baseline life satisfaction measure | At baseline
  Life satisfaction will be assessed using the Satisfaction With Life Scale (SWLS) questionnaire. The scale is composed of 5 items to score with a Likert scale from 1 (strongly disagree) to 5 (strongly agree).
After intervention life satisfaction measure | Immediately after the intervention.
  Life satisfaction after the intervention will be assessed using the Satisfaction With Life Scale (SWLS) questionnaire. The scale is composed of 5 items to score with a Likert scale from 1 (strongly disagree) to 5 (strongly agree).
3 months after intervention life satisfaction measure | 3 months after the intervention ending
  Life satisfaction 3 months after the intervention will be assessed using the Satisfaction With Life Scale (SWLS) questionnaire. The scale is composed of 5 items to score with a Likert scale from 1 (strongly disagree) to 5 (strongly agree).
6 months after intervention life satisfaction measure | 6 months after the intervention ending
  Life satisfaction 6 months after the intervention will be assessed using the Satisfaction With Life Scale (SWLS) questionnaire. The scale is composed of 5 items to score with a Likert scale from 1 (strongly disagree) to 5 (strongly agree).
Baseline self-esteem | At baseline
  Patients' level of self-esteem will be assessed using the Rosenberg Self-Esteem Scale which includes 10 items. Participants will have to score each item with a Likert scale from 1 (strongly disagree) to 4 (strongly agree).
After intervention self-esteem | Immediately after the intervention.
  Patients' level of self-esteem will be assessed after intervention using the Rosenberg Self-Esteem Scale which includes 10 items. Participants will have to score each item with a Likert scale from 1 (strongly disagree) to 4 (strongly agree).
3 months after intervention self-esteem measure | 3 months after the intervention ending
  Patients' level of self-esteem will be assessed 3 months after the intervention using the Rosenberg Self-Esteem Scale which includes 10 items. Participants will have to score each item with a Likert scale from 1 (strongly disagree) to 4 (strongly agree).
6 months after intervention self-esteem measure | 6 months after the intervention ending
  Patients' level of self-esteem will be assessed 6 months after the intervention using the Rosenberg Self-Esteem Scale which includes 10 items. Participants will have to score each item with a Likert scale from 1 (strongly disagree) to 4 (strongly agree).
Baseline anxiety and depression perception measure | At baseline
  Anxiety and depression will be evaluated by the HAD Scale (Hospital Anxiety and Depression Scale). It is composed of 14 items and participants will have to choose one from 4 options to select the affirmation which better corresponds to their perception.
After intervention anxiety and depression perception measure | Immediately after the intervention.
  Anxiety and depression will be evaluated after intervention by the HAD Scale (Hospital Anxiety and Depression Scale). It is composed by 14 items and participants will have to choose one from 4 options to select the affirmation which better corresponds to their perception.
3 months after intervention anxiety and depression perception measure | 3 months after the intervention ending
  Anxiety and depression will be evaluated 3 months after the intervention by the HAD Scale (Hospital Anxiety and Depression Scale). It is composed of 14 items and participants will have to choose one from 4 options to select the affirmation which better corresponds to their perception.
6 months after intervention anxiety and depression perception measure | 6 months after the intervention ending
  Anxiety and depression will be evaluated 6 months after the intervention by the HAD Scale (Hospital Anxiety and Depression Scale). It is composed of 14 items and participants will have to choose one from 4 options to select the affirmation which better corresponds to their perception.
Baseline Shoulder disability perception measure | At baseline
  For the assessment of their perception of disability due to shoulder mobility, the Quick DASH (Disabilities of the Arm, Shoulder and Hand) questionnaire will be used. It is an 11- item self-administered survey referenced over 7 days prior to administration.
After intervention shoulder disability perception measure | Immediately after the intervention.
  For the assessment of their perception of disability due to shoulder mobility, the Quick DASH (Disabilities of the Arm, Shoulder and Hand) questionnaire will be used after the intervention. It is an 11- item self-administered survey referenced over 7 days prior to administration.
3 months after the intervention shoulder disability perception measure | 3 months after the intervention ending
  For the assessment of their perception of disability due to shoulder mobility, the Quick DASH (Disabilities of the Arm, Shoulder and Hand) questionnaire will be used 3 months after the intervention. It is an 11- item self-administered survey referenced over 7 days prior to administration.
6 months after the intervention shoulder disability perception measure | 6 months after the intervention ending
  For the assessment of their perception of disability due to shoulder mobility, the Quick DASH (Disabilities of the Arm, Shoulder and Hand) questionnaire will be used 6 months after the intervention. It is an 11- item self-administered survey referenced over 7 days prior to administration.
Baseline physical activity level measure | At baseline
  The International Physical Activity Questionnaire will be administered to assess the physical activity level of patients before starting the exercise programme. Participants will report the activity performed during the prior 7 days specifying the time spent in each type of physical activity.
After intervention physical activity level measure | Immediately after the intervention.
  The International Physical Activity Questionnaire will be administered to assess the physical activity level of patients after the end of the programme. Participants will report the activity performed during the prior 7 days specifying the time spent in each type of physical activity.
3 months after intervention physical activity level measure | 3 months after the intervention ending
  The International Physical Activity Questionnaire will be administered to assess the physical activity level of patients after 3 months of the end of the programme. Participants will report the activity performed during the prior 7 days specifying the time spent in each type of physical activity.
6 months after intervention physical activity level measure | 6 months after the intervention ending
  The International Physical Activity Questionnaire will be administered to assess the physical activity level of patients after 6 months of the end of the programme. Participants will report the activity performed during the prior 7 days specifying the time spent in each type of physical activity.
Baseline exercise motivation | At baseline
  The existence or not of behavioural change/motivation towards exercise will be assessed before the intervention by using the Behaviour Regulation in Physical Exercise Scale (BREQ-2). The BREQ-2 is a 19 item questionnaire that measures the stages of the self-determination continuum concerning motivation to exercise with a 5 point Likert scale (0=not true for me, 4=very true for me).
After intervention exercise motivation | Immediately after the intervention.
  The existence or not of behavioural change/motivation towards exercise will be assessed after the intervention by using the Behaviour Regulation in Physical Exercise Scale (BREQ-2). The BREQ-2 is a 19 item questionnaire that measures the stages of the self-determination continuum concerning motivation to exercise with a 5 point Likert scale (0=not true for me, 4=very true for me).
3 months after intervention exercise motivation | 3 months after the intervention ending
  The existence or not of behavioural change/motivation towards exercise will be assessed 3 months after the intervention by using the Behaviour Regulation in Physical Exercise Scale (BREQ-2). The BREQ-2 is a 19 item questionnaire that measures the stages of the self-determination continuum concerning motivation to exercise with a 5 point Likert scale (0=not true for me, 4=very true for me).
6 months after intervention exercise motivation | 6 months after the intervention ending
  The existence or not of behavioural change/motivation towards exercise will be assessed 6 months after the intervention by using the Behaviour Regulation in Physical Exercise Scale (BREQ-2). The BREQ-2 is a 19 item questionnaire that measures the stages of the self-determination continuum concerning motivation to exercise with a 5 point Likert scale (0=not true for me, 4=very true for me).
Baseline kinesiophobia | At baseline
  Fear of movement will be measured before intervention by using the Tampa Kinesiophobia Scale. The scale is composed by 17 items that include two subscales, one measures activity avoidance and the other one somatic focus. The total score of the scale range from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia.
After intervention kinesiophobia | Immediately after the intervention.
  Fear of movement will be measured after the intervention by using the Tampa Kinesiophobia Scale. The scale is composed of 17 items that include two subscales, one measures activity avoidance and the other one somatic focus. The total score of the scale range from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia.
3 months after intervention kinesiophobia | 3 months after the intervention ending
  Fear of movement will be measured 3 months after the intervention by using the Tampa Kinesiophobia Scale. The scale is composed of 17 items that include two subscales, one measures activity avoidance and the other one somatic focus. The total score of the scale range from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia.
6 months after intervention kinesiophobia | 6 months after the intervention ending
  Fear of movement will be measured 6 months after the intervention by using the Tampa Kinesiophobia Scale. The scale is composed of 17 items that include two subscales, one measures activity avoidance and the other one somatic focus. The total score of the scale range from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- GOfit, Santander, Cantabria, Spain

REFERENCES:
- [Derived] Lavin-Perez AM, Collado-Mateo D, Hinojo Gonzalez C, de Juan Ferre A, Ruisanchez Villar C, Mayo X, Jimenez A. High-intensity exercise prescription guided by heart rate variability in breast cancer patients: a study protocol for a randomized controlled trial. BMC Sports Sci Med Rehabil. 2023 Mar 8;15(1):28. doi: 10.1186/s13102-023-00634-2. PMID 36890601